CLINICAL TRIAL: NCT05238649
Title: A Randomized, Double Blind, Positive Control Clinical Study to Evaluate the Immunogenicity and Safety of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Against COVID-19 in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines
Brief Title: Immunogenicity and Safety of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine
Acronym: COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ICV-V-01-Booster-A
Record Dates: First submitted 2022-02-10; First posted 2022-02-14 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Vaccines, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- V-01 10 μg (Experimental): 10 μg(0.5ml)/vial, one dose administrated by intramuscular injection
  Interventions: Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine 10μg
- V-01 25 μg (Experimental): 25 μg(0.5ml)/vial, one dose administrated by intramuscular injection
  Interventions: Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine 25μg
- Inactivated vaccine (Active Comparator): 0.5ml/vial, containing 100U inactivated COVID-19 virus antigen. One dose administrated by intramuscular injection
  Interventions: Biological: SARS-Cov-2 Vaccine Inactivated

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine 10μg — The product should be a milky-white suspension for injection. For prevention of SARS-CoV-2 infection.
  Other Names: V-01 10μg
  Arms: V-01 10 μg
Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine 25μg — The product should be a milky-white suspension for injection. For prevention of SARS-CoV-2 infection.
  Other Names: V-01 25μg
  Arms: V-01 25 μg
Biological: SARS-Cov-2 Vaccine Inactivated — The product should be a milky-white suspension for injection. For prevention of SARS-CoV-2 infection.
  Other Names: Inactivated vaccine
  Arms: Inactivated vaccine

SUMMARY:
A Randomized, Double Blind, Positive Control Clinical Study to Evaluate the Immunogenicity and Safety of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Against COVID-19 in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines

DETAILED DESCRIPTION:
This is a Randomized, Double Blind, Positive Control exploratory clinical study. 150 participants aged 18 years and older who have completed the 2 doses of administration of inactive vaccines 6 months (±1 month) ago were enrolled in this study to evaluate the safety and immunogenicity of V-01.

The participants will be enrolled to test group A (V-01 10 μg), test group B (V-01 25 μg) and test group C (inactivated vaccine) by the ratio of 1:1:1. The participants received 1 dose of V-01 or inactivated vaccine base on the group.

The random stratification factor is age (18-59 years old vs. ≥ 60 years old).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged 18 years and older who have completed the second dose of 2-dose regimen of SARS-CoV-2 Inactivated Vaccine in the past 6 (±1) months;
2. Voluntarily participate in the study and sign the informed consent form, who can provide valid ID and follow the study protocol requirement;
3. In the past 14 days, no history of high or medium risk of the epidemic, overseas travel history or residence history; no history of contact with confirmed, asymptomatic or suspected COVID-19 cases; no history of contact with the persons from high- and medium-risk epidemic areas or contact patients with fever or respiratory symptoms; and those who are not in isolation period.
4. Males of reproductive potential and females of childbearing potential voluntarily agree to take effective and acceptable contraceptive methods from the signing of informed consent form to 3 months after vaccination.

Exclusion Criteria:

1. Confirmed COVID-19 cases, or positive for SARS-CoV-2 test by RT-PCR. 2. History of previous SARS infection. 3. History of severe allergy to any vaccine or any ingredient of the vaccine including aluminum adjuvant, e.g., anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), dyspnea, angioedema, etc.

4. People who currently suffer from the following diseases:

1. Symptoms related to acute respiratory infections (such as: sneezing, nasal congestion, runny nose, cough, sore throat, loss of taste, chills, shortness of breath, etc.)
2. Patients with thrombocytopenia, any coagulation dysfunction, or receive anticoagulant treatment, etc.
3. Patients with congenital or acquired angioedema/neuroedema;
4. A history of congenital or acquired immunodeficiency or autoimmune disease (except for mild psoriasis, controllable autoimmune thyroid disease, vitiligo, or stable celiac disease that does not require immunosuppressive or immunomodulatory therapy); no spleen , or history of spleen surgery, history of trauma, or treatment with immunomodulators within 6 months, such as: glucocorticoid with the dose causing immunosuppressive (dose reference: equivalent to prednisone 20mg/day, more than one week); or monoclonal antibody ; or thymosin; or interferon, etc.; but local medication (such as ointment, eye drops, inhalation or nasal spray) is allowed.
5. Patients with active tuberculosis, viral hepatitis, human immunodeficiency virus or syphilis infection.
6. Patients with acute diseases, or acute attacks of chronic diseases, or uncontrolled severe chronic diseases: history of chronic respiratory diseases (including moderate to severe asthma, COPD, pulmonary fibrosis), hypertension that cannot be controlled by drugs (systolic blood pressure ≥150mmHg) And/or diastolic blood pressure ≥100mmHg), history of severe cardiovascular disease (including heart failure, coronary artery disease, cardiomyopathy), history of chronic kidney disease, history of cancer (except for basal cell carcinoma), diabetes (unsatisfied blood sugar control or diabetes related serious complications).

5. Received inactivated vaccines or any subunit vaccines within 14 days before the vaccination and attenuated live vaccine within 28 days before the vaccination.

6. Injection of immunoglobulin and/or other blood products within 3 months before the administration of study vaccine; or with the plan to use such product within 6 month after immunization.

7. Pregnant (including positive urine pregnancy test for women of childbearing age) or breastfeeding women. Or women or their partners who have a pregnancy plan within 3 months after the trial vaccination.

8. Have participated in or are participating in other COVID-19 related clinical trials, or are participating in other drug clinical trials; 9. Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-28 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers of SARS-CoV-2 neutralizing antibodies | 28 days after booster immunization
  The Geometric Mean Titers of SARS-CoV-2 neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ligong Lu, Dr., Principal Investigator — Zhuhai People's Hospital Medical Group
Locations (1):
- Zhuhai Peoples' Hospital Medical Group, Zhuhai, Guangdong, China